CLINICAL TRIAL: NCT02743442
Title: Da Vinci Transoral Robotic-assisted Surgery of Pituitary Gland
Acronym: ROBOPHYSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCT-2015-043
Record Dates: First submitted 2016-04-04; First posted 2016-04-19 (Estimated); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Pituitary Neoplasms
MeSH Terms: conditions — Pituitary Neoplasms

ARMS (1):
- Transoral surgery (Experimental)
  Interventions: Device: da Vinci® Si™

INTERVENTIONS:
Device: da Vinci® Si™

SUMMARY:
Over the past 30 years, endoscopic transnasal techniques have gained a major interest, and anatomic limits have been widened in order to extend neurosurgical applications. For many years, robotic-assisted surgery using the da Vinci system (Intuitive Surgical Inc, Sunnyvale, California, USA) has been greatly developed, especially in urology and gynecology.

Robotic-assisted surgery has been performed for pharyngeal and laryngeal cancers in a minimally invasive perspective.

A robot-assisted preliminary series demonstrated the ability to approach the sella via oral approach without traumatic injury of nasal or oral cavity. Transoral approach avoids the complications of the endonasal resection: synechia, rhinitis sicca anterior, primary and secondary atrophican rhinitis, and empty nose syndrome.

The investigators recently published a cadaveric study of transoral robotic-assisted skull base surgery to approach the sella turcica (Neurosurgical Rev. 2014; 37:609-17).

In this study, the investigators will propose a new minimally invasive technique of pituitary surgery by transoral approach assisted by the da Vinci robot in patients with pituitary adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Pituitary adenoma with a surgical indication : visual compression and chiasmal syndrome, intracranial hypertension , hormonal syndrome (hypopituitarism and hypersecretion ) , failure of medicamentous treatments for prolactinoma
* No pituitary apoplexy (requiring emergency surgery)
* Spontaneous oral opening greater than 35 mm

Exclusion Criteria:

* Insufficient buccal opening
* Intercurrent pathology of oropharyngeal and nasopharyngeal
* Complicated forms of adenoma pituitary adenoma (invasive adenoma)
* Hemostasis disorder
* Phlebitis or active pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Transoral Surgery: da Vinci® Si™ single arm
Period: Overall Study
Arm/Group | Transoral Surgery
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients were included between 2016 and 2018. The median age was 48 (minimum: 22 years, maximum: 69 years).
  The median follow-up (time between the inclusion date and the end of the follow-up) was 6 months and 10 days.
Groups:
- Transoral Surgery: The study is a single arm : all patients were treated with da Vinci surgical procedure.
Arm/Group | Transoral Surgery
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.25 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  France | 8
Size of the lesion before surgery [Mean (Standard Deviation); unit: millimeters] | 30.75 (6.14)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Operated Via da Vinci Robot
Description: Number of patients in which the entire sella turcica (including its anterior face) is seen during surgery and reached by the robotic arms
Time Frame: 1 day
Population: Among the 8 patients enrolled in this study, 7 were operated using the Vinci robot. The surgery was canceled for one patient with acute coronary syndrome (a serious adverse event not related to the study).
Measure: Number; unit: participants
Groups:
- Transoral Surgery: Surgery of the pituitary adenoma via a transoral approach assisted by the da Vinci® Si™ robot
Arm/Group | Transoral Surgery
Number analyzed (Participants) | 7
participants | 7

2. Secondary Outcome: Duration of Surgery
Description: Total duration of surgery: installation, mucosal time, sphenoidal time, resection and closure
Time Frame: 3 hours
Reporting Status: Not Posted

3. Secondary Outcome: Number of Severe Adverse Events
Description: An adverse event occurring after the procedure is serious if it causes death, endangers the life of the person who is suitable for research, requires or prolongs hospitalization, causes a significant handicap, results in a congenital malformation, or is considered medically significant.
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization after surgery
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definition of an adverse event: any harmful manifestation occurring in a person who is amenable to research involving the human person, whether or not the event is related to the research or product to which the research relates.
  Definition of a serious adverse event: any adverse event that causes death, is life-threatening, requires hospitalization or prolongation, causes disability, results in a congenital malformation, and any event considered medically significant.
Arm/Group | Transoral Surgery
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transoral Surgery (N=8)
Complication of neurological intervention (Surgical and medical procedures) | 1 (1) — Rhinorrhea with cerebrospinal fluid
Injury, poisoning and complications of interventions (Surgical and medical procedures) | 2 (2) — Resumption of surgery
Injuries and complications related to an intervention (Cardiac disorders) | 1 (1) — Acute coronary syndrome during anesthesia (surgery of excision of the adenoma canceled)
Stroke (Vascular disorders) | 1 (1) — Stroke post surgical revision
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transoral Surgery (N=8)
Diabetes insipidus (Endocrine disorders) | 3 (3) — polyuro-polydipsic syndrome
Headaches (Nervous system disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 2 (2)
Laryngeal pain (General disorders) | 3 (3)
Visual trouble (Eye disorders) | 3 (3)
Asthenia (General disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Post-lumbar puncture syndrome (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumocephalus (Nervous system disorders) | 1 (1)
Corticotropin deficiency (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Paralysis of the nerve III (Eye disorders) | 1 (1)
Pain at the incision site (Injury, poisoning and procedural complications) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02743442/Prot_SAP_000.pdf